CLINICAL TRIAL: NCT04035642
Title: Phase II Study of Single-Dose Image-Guided Radiotherapy (SDRT) With Urethral Sparing for Localized Prostate Cancer
Brief Title: Phase II Study of Single-Dose Image-Guided Radiotherapy (SDRT) for Prostate Cancer
Acronym: PROSINT II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Carlo Greco, MD, Principal Investigator, Fundacao Champalimaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROSINT II
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGRT 24 Gy Single dose (Experimental): Patients will be treated using image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. Patients will be treated with a single fraction at a prescription dose of 24 Gy.
  Interventions: Radiation: IGRT 24 Gy Single dose; Procedure: Image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT); Device: Rectal balloon with air filling; Device: Urethral catheter loaded with beacon transponders

INTERVENTIONS:
Radiation: IGRT 24 Gy Single dose — Previously untreated patients with prostate cancer will be treated with 24Gy in in one session.
Procedure: Image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) — Patients enrolled in the study will undergo IGRT-VMAT with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility.
Device: Rectal balloon with air filling — A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility.
Device: Urethral catheter loaded with beacon transponders — A urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking.

SUMMARY:
The present study evaluates clinical outcomes and treatment-related toxicity following definitive ultra-high single dose external beam radiotherapy delivered to patients with low- or intermediate-risk adenocarcinoma of the prostate. Modern computer-driven technology enables the implementation of ultra-high Single-Dose Image-Guided Radiotherapy (SD-IGRT) safely.

Prostate cancer patients classified according to the current National Comprehensive Cancer Network (NCCN) guidelines as low or intermediate risk (biopsy Gleason score of ≤7 and/or Prostate Specific Antigen (PSA) level ≤20 ng/mL and/or Stage T1, T2a, T2b or T2c) are eligible for this study.

Patients will undergo SD-IGRT with volumetric intensity-modulated arc radiotherapy (VMAT) with state-of-the-art treatment-planning and quality assurance procedures. Emphasis is placed on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with low- or intermediate-risk prostate cancer will receive 24 Gy in a single-dose.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus, though not exclusively, on urinary, rectal and sexual functions and will be assessed through validated EPIC questionnaires. Serum PSA values will be drawn on the same schedule as clinical follow-up. A multi-parametric MRI will be performed at baseline, and at 6, 12 and 24 months following intervention. The study will be continuously monitored for a minimum of 5 years.

DETAILED DESCRIPTION:
The present phase II study evaluates the clinical outcomes and potential treatment-related toxicity following definitive ultra-high dose single fraction external beam radiation therapy (SDRT) in patients with localized adenocarcinoma of the prostate. A large body of data suggests that extreme hypofractionated radiation schedules, which employ ultra-high dose per fraction (≥7 Gy) in a small number of fractions (≤5), appear equal or superior to conventionally-fractionated (1.8-2.0 Gy/fraction) and moderately hypo-fractionated schemes (2.5-3.5 Gy/fraction) in terms of both tumor control and toxicity profiles. Modern computer-driven technology enables the implementation of ultra-high hypofractionated Image-Guided Radiotherapy (IGRT) safely. The Radiation Oncology team at Champalimaud Centre for the Unknown has been engaged in a large phase II study (HYPO) of extreme hypofractionation (9Gyx5) which accrued over 200 cases and, with a median follow-up of over 3 years, showed the safety and efficacy of this approach. The feasibility of SDRT in localized prostate cancer has been tested by the in a randomized phase II trial (PROSINT) comparing extreme hypofractionation as per the HYPO trial regimen vs. a single dose of 24Gy. While the long-term results of this study are still pending, its toxicity profile in both arms has been extremely good with no G3 adverse events at 2 years and superimposable biochemical response between the two regimens. Taken together, these observations provide the basis for the prospective clinical studies proposed herein.

Patients enrolled in the study will undergo image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with low and intermediate risk (NCCN criteria) localized prostate cancer will be treated with 24 Gy SDRT.

Patients will be followed at one and three months post-treatment, every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus, though not exclusively, on urinary, rectal and sexual functions and will be assessed through validated EPIC questionnaires. Serum PSA values will be drawn on the same schedule as clinical follow-up. A multiparametric MRI will be performed at baseline, and at 6, 12 and 24 months following intervention. The study will be continuously monitored for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form;
* Histologic confirmation of adenocarcinoma of the prostate by biopsy;
* Up to 6 months of previous hormonal therapy is allowed (but not required)
* PSA ≤ 20 prior to hormone therapy (if given);
* Biopsy Gleason score ≤ 7
* No direct evidence of regional or distant metastases after appropriate staging studies
* Age ≥ 18
* Performance Status 0-2
* American Urological Association (AUA) score must be ≤ 20 (alpha blockers allowed)
* Computerized Tomography (CT) or Ultrasound-based volume estimation of prostate gland ≤ 100 grams

Exclusion Criteria:

* Positive lymph nodes or metastatic disease from prostate cancer on imaging studies
* Prior invasive malignancy unless disease free for a minimum of 3 years
* MRI evidence of radiographic T3, T4 or N1 disease
* Tumour Clinical stage T3 or T4 on MRI
* PSA > 20 ng/mL
* Gleason score > 7
* Previous pelvic radiotherapy
* Previous surgery for prostate cancer
* Recent transurethral resection of the prostate (TURP) (less than 3 months)
* Previous hormonal therapy given for more than 6 months prior to therapy
* Previous significant urinary obstructive symptoms;
* Significant psychiatric illness
* Ultrasound or CT estimate of prostate volume > 100 grams
* Severe, active co-morbidity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0 | 5 years
  Comparison of treatment related adverse events as measured by Common Toxicity Criteria for Adverse Effects v4.0 over a 5 year time frame.
Concentration of serum PSA | 5 years
Changes in PSA biochemical parameter measurements (Phoenix Definition). | 5 years

SECONDARY OUTCOMES:
Assessment of imaging response based on multi-parametric MRI | 24 months
Expanded Prostate Cancer Index Composite (EPIC) Questionnaire to measure quality of life | 5 years
  Quality of life is measured on a scale of 0 to 100, with higher scores representing a higher quality of life.
International Index of Erectile Function (IIEF) Questionnaire assess sexual function | 5 years
  Sexual function is measured on a scale of 0 to 75, with higher scores representing higher sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, MD, Principal Investigator — Fundacao Champalimaud
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal